CLINICAL TRIAL: NCT02923284
Title: Nanotech Biomarkers For Renal Cancer Intervention: Clinical Validation & Utility
Brief Title: NANOTECH RCC Biomarkers
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 201601082; 5R01CA141521 (NIH)
Record Dates: First submitted 2016-09-07; First posted 2016-10-04 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Renal Cell Carcinoma; Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples will be retained with a study-specific code that links the samples to data collected from the electronic medical record.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Imaged renal mass cohort: Subjects undergoing surgery for an kidney tumor identified radiologically.
- control cohort: Subjects undergoing surgery for any kind of cancer other than kidney.

SUMMARY:
The incidence of renal cell carcinoma (RCC or kidney cancer) in men exceeds that of pancreatic cancer or leukemia. In women, the incidence of RCC is similar to that of leukemia, ovarian, or pancreatic cancer; thus, RCC is significant health issue. This study focuses on identifying specific molecules [biomarkers] of RCC that can be used to develop a reliable low-cost screening method at the point of service. If successful, our method would provide a diagnostic test to distinguish benign kidney masses from malignant ones, eliminating the need to surgically remove a kidney with a benign tumor.

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years of age and older undergoing surgery. Patient samples are divided into 2 groups based on their surgery: Patients with an imaged renal mass, encompassing about 300 patients/year (about 1200 total) of both malignant (about 80-85% of time) and benign (about 15-20% of time), and patients with non-kidney cancers, encompassing about 6,000 patients/year (about 24,000 total),

Exclusion Criteria:

Age <18 years and prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are 18 years of age and older and undergoing planned surgical procedure for removal of an imaged renal mass will be consented in the Center for Preoperative Assessment and Planning (CPAP), the holding area on the day of surgery, and the holding area of radiology. A urine sample will be collected from subject following informed consent. Additionally, discarded urine samples will be collected from the BJH Chemistry Labs from patients admitted for surgery for non-kidney cancer as a comparator group.
Sampling Method: Non-Probability Sample
Enrollment: 407 (Actual)
Dates: Start 2016-08; Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Urine AQP1 | 28 days
  Assay results will be compared to the pathology report for the excised renal mass and the ICD10 codes.
PLIN2 concentration | 28 days
  Assay results will be compared to the pathology report for the excised renal mass and the ICD10 codes.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremiah Morrissey, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University St Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No